CLINICAL TRIAL: NCT05048160
Title: Phase I/II Clinical Trial of 6MW3211 Injection to Evaluate Safety, Tolerability, PK/PD, Immunogenicity and Preliminary Efficacy in Subjects With Advanced Malignant Neoplasm.(Only Phase I Has Been Submitted to US FDA)
Brief Title: A Clinical Study of 6MW3211 Injection in the Treatment of Advanced Malignant Neoplasm
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6MW3211-2021-CP101
Record Dates: First submitted 2021-08-31; First posted 2021-09-17 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Advanced Malignant Neoplasm
MeSH Terms: interventions — Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 6MW3211 (Experimental): * Dosage form: injection
  * Specification: 240 mg / 8 ml/Vial
  Interventions: Drug: Intravenous Infusion

INTERVENTIONS:
Drug: Intravenous Infusion — Dose-limiting toxicity (DLT) are assessed during the first 3 weeks (21 days) after initial administration. Then, the intended dosing frequency is every 2 weeks (Q2W).

SUMMARY:
This study is a single arm, non-randomized, open label, multiple doses phase I/II international, multicenter clinical trial to evaluate safety, tolerability, PK/PD, immunogenicity and preliminary efficacy in subjects with advanced malignant neoplasm. The study is consisted of two stages: dose escalation and clinical expansion.

Only Phase I has been submitted to US FDA,and the protocol number is still the same as 6MW3211-2021-CP101.The US title is : A Phase 1, First-in-Human (FIH), Multicenter, Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of 6MW3211 in Patients with Advanced Malignancies .

DETAILED DESCRIPTION:
Six cohorts are included in dose escalation stage, at doses of 0.3~45 mg/kg, respectively. Safety, tolerability, and dose-limiting toxicity (DLT) are assessed during the first 3 weeks (21 days) after initial administration. Then, the intended dosing frequency is every 2 weeks (Q2W), IV.

From the first study drug administration, some dosing cycles will be observed for phase I, initial tumor efficacy assessments will be performed at week 7, after that tumor efficacy assessment will be carry out for every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1. Men or women, age ≥18.
* 2.Subjects with advanced malignancy histopathologically and/or cytologically, with at least one evaluable tumor lesion.
* 3.ECOG PS is 0 or 1.
* 4.Survival expectation of at least 3 months.
* 5.Adequate organs and hematopoietic functions
* 6.Voluntarily signing of informed consent

Exclusion Criteria:

* 1.Subjects with brain metastases of clinically active central nervous system (CNS).
* 2.Subjects that require to take anticoagulants and/or aspirin.
* 3.Blood transfusion within 2 weeks prior to the first administration of study treatment.
* 4.Inadequately controlled body cavity effusions.
* 5.Subjects with active, or have a history and possible recurrence of autoimmune diseases .
* 6.Have uncontrolled systemic diseases.
* 7.Subjects who had received anticancer therapy or radiotherapy within 4 weeks or 5 half-lives (whichever is shorter) before enrollment.
* 8.Subjects are known to have previously experienced severe allergic reactions to large molecular protein formulations/monoclonal antibodies.
* 9.Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
AEs | Up to 28 days post last dose
  All the adverse events
ORR | 1 Year
  Objective Response Rate
DOR | 1 Year
  Duration of Remission
PFS | 1 Year
  Progression-Free Survival
DCR | 1 Year
  Disease Control Rate
OS | 1 Year
  Overall Survival

SECONDARY OUTCOMES:
PK Parameters | 1 Year
  The area under the curve (AUC)
PK Parameters | 1 Year
  Maximum concentration(Cmax)
PK Parameters | 1 Year
  Time at which maximum concentration(Tmax)
PK Parameters | 1 Year
  The half life(T1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Professor, Principal Investigator — Fudan University Cancer Hospital of China
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No